CLINICAL TRIAL: NCT06238388
Title: A Phase I Clinical Trial Exploring the Metabolic and Excretion Characteristics of HSK21542 Injection in Maintenance Hemodialysis Patients
Brief Title: Metabolism and Excretory of HSK21542 in Maintenance Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK21542-105
Record Dates: First submitted 2024-01-21; First posted 2024-02-02 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 0.8 μg/kg HSK21542 Injection (Experimental): 0.8 μg/kg HSK21542 Injection
  Interventions: Drug: HSK21542 Injection

INTERVENTIONS:
Drug: HSK21542 Injection — A single intravenous dose of 0.8 μg/kg HSK21542 in boluses after D1 dialysis completed.

SUMMARY:
This is a single-center, nonrandomized, and open design study to investigate metabolism and excretion of HSK21542 in maintenance hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to sign an informed consent form, fully understand the objectives and purposes of the study, and are willing to comply with the study protocol before any of the study-related procedures start.
2. Age ≥18 years old, Male or female;
3. Patients with end-stage renal diseases who receive hemodialysis (including hemodiafiltration) 3 times in a week prior to screening for at least 3 months;
4. Dry weight is 40.0-135.0 kg (inclusive) during the screening period;
5. Patients with at least two occurrences of single-compartment urea clearance (sp Kt/V) ≥ 1.2, or at least two occurrences of urea reduction ratio (URR) ≥ 65%, or one occurrence of sp Kt/V ≥ 1.2 and one occurrence of URR ≥ 65% on different days of dialysis within 6 months before administration;
6. Female of childbearing age or Male must agree to adopt efficient contraceptive measures in sexual intercourse during the study period and within 3 months after the last administration; Menopausal female subjects should have had menopause at least one year or should have had permanent sterilization (e.g., fallopian tube occlusion, hysterectomy, bilateral salpingectomy).

Exclusion Criteria:

1. Expected to undergo kidney transplantation and/or parathyroidectomy during the study;
2. History of allergy to opioids, such as urticaria (Note: adverse effects related to opioid use, such as constipation and nausea, are not included as the exclusion criteria in this study);
3. Used opioids within 7 days before screening, or unable to avoid the use of opioids other than the investigational product during the study;
4. Participated in any clinical trial of other drug or medical device within 1 month before screening (received study medication or treated by the medical device in the clinical trial);
5. Used blood perfusion during the screening period or expected study period;
6. Blood pressure of upper limbs in the supine position at screening: systolic blood pressure < 90 mmHg, or diastolic blood pressure < 60 mmHg, or systolic blood pressure > 180 mmHg, or diastolic blood pressure > 110 mmHg;
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)≥ 2.5 × upper limit of normal (ULN), or total bilirubin ≥ 2 × upper limit of normal (ULN) at screening;
8. Blood sodium > 155 mmol/L at screening;
9. Blood donation (or loss) ≥ 400 mL within the first 3 months of screening or Hemoglobin < 80 g/L at screening;
10. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody;
11. Females who are pregnant or breastfeeding;
12. Smoking an average of more than 5 cigarettes per day within the first 3 months of screening, or not stopping the use of any tobacco products during the trial period;
13. Any physiological or psychological diseases or conditions that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial, as judged by the study physician, including but not limited to:

    1. Known or suspected alcohol, anesthetic, or other substance abuse or drug dependence history within the first 12 months of screening; Baseline urine drug screening (if any) or positive alcohol breath test;
    2. severe systolic or diastolic heart failure within the first 6 months of screening (e.g. NYHA grade IV congestive heart failure (NYHA heart function grading criteria can be found in Appendix 3) ;
    3. Severe mental illness or cognitive impairment (e.g., dementia);
    4. Any other relevant acute or chronic neurological and psychiatric diseases (e.g., encephalopathy, coma, delirium) within 3 months before screening And the researchers believe it is not suitable for enrollment;
    5. Patients with malignant tumors, but not including: curable cervical carcinoma in situ, skin basal cell carcinoma, or squamous cell carcinoma, or any other tumor that has been cured (with no evidence of disease recurrence within 5 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery of unchanged drug (Ae) | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in urine, feces, and dialysate
Cumulative recovery fraction of unchanged drug (Fe) | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in urine, feces, and dialysate
Plasma clearance | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in urine, feces, and dialysate
Cmax | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in plasma
AUC(0-t) | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in plasma
AUC(0-∞) | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in plasma
Tmax | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in plasma
t1/2 | From the start of administration to 168 hours after administration
  The pharmacokinetic parameters of HSK21542 in plasma

SECONDARY OUTCOMES:
The main metabolites of HSK21542 | From the start of administration to 168 hours after administration
  The main metabolites of HSK21542 in plasma, urine, feces, and dialysate
Adverse events (AEs) | From after administration to the end of telephone follow-up
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No